CLINICAL TRIAL: NCT01472172
Title: Pleural Cryobiopsies During Semirigid Thoracoscopy: A New Technique
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Principal Investigator, Aleš Rozman, Head of endoscopy department, The University Clinic of Pulmonary and Allergic Diseases Golnik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Endo-0002
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Pleural Effusion; Pleural Diseases
Keywords: Flex-rigid pleuroscopy; cryobiopsy; pleural biopsy; pleural effusion; safety; thoracoscopy
MeSH Terms: conditions — Pleural Effusion; Pleural Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryobiopsy (Experimental): Biopsies will be obtained by flexible autoclavable cryoprobe 20416-032 (Erbokryo CA, ERBE, Germany) with 2.4 mm in diameter. The tip of the probe is cooled to -890C with nitrous oxide within seconds after footswitch activation. The biopsy sample will by extracted by gently pulling of the probe.
  Interventions: Device: Cryobiopsy (Autoclavable cryoprobe 20416-032)

INTERVENTIONS:
Device: Cryobiopsy (Autoclavable cryoprobe 20416-032) — The tip of the cryoprobe will be attached to suspicious part of parietal pleura and activated by footswitch for 3 seconds. The frozen tissue is going to be extracted by gently pulling of the probe. The probe with the attached biopsy sample is going to be removed together with the thoracoscope through trocar. The biopsy sample will be released from the probe by thawing in the saline.
  Other Names: Autoclavable cryoprobe 20416-032 (ERBE, Germany)

SUMMARY:
The purpose of this study is to determine feasibility of pleural biopsies with the cryoprobe during semirigid thoracoscopy. The secondary aim is to evaluate safety with focus on bleeding intensity.

DETAILED DESCRIPTION:
The primary aim of this study is to determine feasibility of pleural biopsies with the cryoprobe during semirigid thoracoscopy. We will assess size, morphological features, immunohistochemistry and diagnostic yield as measures of the quality of the samples. The secondary aim is to evaluate safety with focus on bleeding intensity.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years old
* Unilateral pleural effusion of unknown origin
* Pleural irregularities suspicious for pleural malignancy
* Referral for thoracoscopy after less invasive means of diagnosis had failed

Exclusion Criteria:

* Uncontrolled bleeding tendency
* Unstable cardiovascular status
* Severe heart failure
* ECOG performance status 4
* Persistent hypoxemia after evacuation of pleural fluid
* Pleural symphisis, fibrothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number / percent of patients with useful pleural biopsy sample, obtained by cryoprobe | 12 months
  To determine, wheather cryobiopsy specimen can be obtained in each patient
Size of biopsy samples | 12 months
  Size of the biopsy specimens in mm2
Quality of the sample | 12 months
  Interpretability of biopsy specimens in histopathology terms: 1. easily interpretable (enough tissue with all elements required for diagnosis) 2. interpretable with some difficulty (less tissue or diagnostic elements - diagnosis less reliable) 3. interpretable with great difficulty (little tissue or scarce diagnostic elements - low reliability of diagnosis) 4. non-interpretable (diagnosis not possible)
  Assessment of biopsy-related artifacts by describing the amount of unaltered tissue in quartiles

SECONDARY OUTCOMES:
Bleeding | 1 month
  Number of patients with a certain degree of bleeding from biopsy site, described as:
  1 = slight, self-limited, 2 = moderate, requiring electrocautery intervention, 3 = severe, requiring interruption of the procedure, chest tube drainage and intravenous fluid resusucitation.

CONTACTS AND LOCATIONS:
Overall Officials: Ales Rozman, MD, Principal Investigator — University Clinic Golnik
Locations (1):
- University Clinic Golnik, Golnik, Golnik, Slovenia